CLINICAL TRIAL: NCT05122572
Title: An Open-label Clinical Study to Evaluate the Safety and Efficacy of Intravenous With and Without Intratumoral Oncolytic Virus Injection (RT-01) Combined With or Without Immune Checkpoint Inhibitors (Nivolumab) in the Treatment of Patients With Advanced Solid Tumors
Brief Title: RT-01 Monotherapy and in Combination With Nivolumab in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuxi People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LWY21076C2
Record Dates: First submitted 2021-11-02; First posted 2021-11-16 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2021-11

CONDITIONS: Advanced Solid Tumor
Keywords: RT-01; Oncolytic Virus Injection; Inmmune Checkpoint Inhibitors; Intravenous Injection; Intratumoral Injection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intravenous Injection (Experimental): Intravenous with or without Intratumoral RT-01 in the treatment of patients with advanced solid tumors combined with or without Nivolumab in the treatment of patients with advanced solid tumors
  Interventions: Biological: Oncolytic Virus Injection (RT-01）

INTERVENTIONS:
Biological: Oncolytic Virus Injection (RT-01） — Intravenous injection of RT-01 with or without Nivolumab

SUMMARY:
This is a single-arm, open-lable study to determine the safety, tolerability and preliminary efficacy of oncolytic virus injection (RT-01) combined with or without immune checkpoint inhibitors (Nivolumab) in the treatment of patients with advanced solid tumors.

DETAILED DESCRIPTION:
To evaluate the safety, tolerability, efficacy, immunoreactivity, immunogenicity, pharmacokinetics and virus shedding of RT-01 injection given via Intravenous with or without Intratumoral administration combined with immune checkpoint inhibitors Nivolumab in the treatment of patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years;
* Have a histopathologically or cytologically confirmed dagnosis of advanced solid tumors and no existing options are felt to provide clinical benefit;
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) (non-nodal lesions with longest diameter ≥ 10 mm, or nodal lesions with short diameter ≥ 15 mm);
* ECOG score of 0 ~ 2;
* Adequate bone marrow, hepatic and renal and cardiovascular function;
* Women of childbearing age who have a negative pregnancy test within 7 days before treatment. Female patients of childbearing age, and male patients with partners of childbearing age must agree to use at least one medically recognized contraceptive method during study treatment and within at least 6 months after the last dose of investigational drug;
* Ability to provide written informed consent.

Exclusion Criteria:

* Subjects with known brain metastasis and/or clinically history tumor brain of metastasis；
* Subjects who have received anti-tumor therapy such as chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy, etc within 4 weeks；
* Subjects who have participate in another interventional study while receiving study IP within 4 weeks；
* Subjects who have had major surgery ≤ 4 weeks of dosing；
* Patients in any condition requiring systemic treatment with corticosteroids (prednisone > 10 mg/day or equivalent of the similar drug) or other immunosuppressive agents within 14 days prior to investigational drug administration, but currently or previously treated with any of the following steroid regimens, were included:
* Topical, ophthalmic, intra-articular, intranasal, or inhaled corticosteroids with minimal systemic absorption;
* Prophylactic short-term (≤ 7 days) use of corticosteroids (e.g., allergy to contrast media) or for the treatment of non-autoimmune diseases (e.g., delayed hypersensitivity caused by contact allergens)；
* Subjects received live vaccines within 7 days of initiation of study treatment；
* Subjects with adverse reactions caused by previous anti-tumor treatment not recovered to (CTCAE 5.0) grade 1 (except alopecia)；
* Subjects who have any active infection；
* Subjects with known positive history of human immunodeficiency virus (HIV) test or known acquired immunodeficiency syndrome (AIDS)；
* Subjects who have active hepatitis；
* Subjects who have serious cardiovascular system disorders history；
* Subjects with active autoimmune diseases or history of autoimmune diseases that may relapse；
* Subjects having any serious uncontrolled disease or in other conditions that would preclude them from receiving study treatment and are considered unsuitable for this study in the opinion of the investigator；
* Subjects in other conditions that are considered unsuitable for this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | Up to 28 days
  Graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Defined as the highest safety-tolerated dose level where at most one patient out of six experiences dose limiting toxicities (DLT) with the next higher dose level having at least 2 of 6 patients who have experienced DLT.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 6 months
  Graded according to the NCI CTCAE version 5.0.
Overall response rate (ORR) | Up to 6 months
  Proportion of patients in the analysis population who have complete response (CR) or partial response (PR) based on RECIST v1.1 imaging.
Disease Control Rate (DCR) | Up to 6 months
  Proportion of patients in the analysis population who have complete response (CR), partial response (PR) or stable disease (SD) based on RECIST v1.1 imaging.
Overall Survival (OS) | Up to 6 months
  Survival time is defined as the time from registration to death due to any cause.
Progression Free Survival (PFS) | Up to 6 months
  Progression-free survival is defined as the time from registration to the earliest date documentation of disease progression or death due to any cause.
Viral replication and shedding in blood, urine and buccal swabs | Up to 6 months
  Assessed via quantitative reverse transcriptase polymerase chain reaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuxi People's Hospital, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No